CLINICAL TRIAL: NCT06447584
Title: Clinical Spectrum and Outcome of Poisoning in Children Admitted to the Pediatric Emergency and Intensive Care Units at Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Asaad Saber, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-24-5-2024-09MS
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Acute Poisoning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute poisoning is a major health problem that leads to emergent hospital admission.It has become the main factor that harms children and leads to disability and death of children. Also, it is still a serious issue in developing countries where it represents a common cause of emergency department presentation and admission. Acute poisoning can be divided into two categories (accidental and intentional),accidental poisoning is common in children under five years, whereas intentional poisoning is more common in adolescents, WHO estimated that, in 2016, accidental poisoning caused 106,683 deaths and the loss of 6.3 million years of healthy life.

A study in Romania showed that intentional poisoning is the most common cause of poisoning among teenagers. Females are more vulnerable to suicidal or intentional poisoning than males. Medications, alcohol, and substance abuse are common poisoning agents among teenagers , another study at tertiary Indian hospital, pesticides, pharmaceutical drugs, and household products were the most common types of acute poisoning. Pesticides were reported as a cause of intentional and accidental poisoning. In agricultural areas, people were poisoned accidentally by pesticides that may be used for suicidal attempts because of their availability. Pharmaceutical drugs are also used for intentional poisoning due to the availability of street drugs and over-the-counter medications. Accidental poisoning by household products were observed in children and the most common products are hydrocarbon and naphthalene In Egypt acute poisoning represents a significant proportion of emergency visits of children and young people. This labors a burden on healthcare, society and economy and thus, it drain-s resources and multiplies workload . In fact, it is a preventable cause of morbidity and mortality. Children poisoning is a result of multiple risk factors including social, demographic, and industrial factors. Insufficient public awareness, easy accessibility to poison, negligence of caregivers, technological and industrial advances and even the nature of the environment are of the main causes.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to pediatric emergency and intensive care units with claim or suspected to have acute poisoning aged from 1 month Up to 18 years old.

Exclusion Criteria:

* Children with chronic poisoning
* no clear history or clinical picture of definite toxic poison
* incomplete clinical data

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients admitted to pediatric emergency and intensive care units with claim or suspected to have acute poisoning aged from 1 month Up to 18 years old.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Recovery Time of acute poisoning | 1 year
  Full Recovery with appropriate and timely medical intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Jesslin J, Adepu R, Churi S. Assessment of prevalence and mortality incidences due to poisoning in a South Indian tertiary care teaching hospital. Indian J Pharm Sci. 2010 Sep;72(5):587-91. doi: 10.4103/0250-474X.78525. PMID 21694990
- [Background] Ballesteros MF, Williams DD, Mack KA, Simon TR, Sleet DA. The Epidemiology of Unintentional and Violence-Related Injury Morbidity and Mortality among Children and Adolescents in the United States. Int J Environ Res Public Health. 2018 Mar 28;15(4):616. doi: 10.3390/ijerph15040616. PMID 29597289
- [Background] Heron M. Deaths: Leading Causes for 2015. Natl Vital Stat Rep. 2017 Nov;66(5):1-76. PMID 29235984
- [Background] Abdel Baseer KA, Gad EF, Abdel Raheem YF. Clinical profile and outcome of acute organophosphate poisoning in children of Upper Egypt: a cross-sectional study. BMC Pediatr. 2021 Feb 26;21(1):98. doi: 10.1186/s12887-021-02563-w. PMID 33637060